CLINICAL TRIAL: NCT02403687
Title: Prospective Analgesic Compound Efficacy (PACE) Study
Acronym: PACE
Status: Completed | Type: Observational
Sponsor: Express Specialty Pharmacy (Other)
Responsible Party: Principal Investigator, Kate McLellan, Study Director, Express Specialty Pharmacy
Other Study IDs: 1960fp-expr-201501
Record Dates: First submitted 2015-03-05; First posted 2015-03-31 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Arthritis; Tendonitis; Gout; Radiculopathy; Muscle Spasms; Synovitis; Migraine; Headache
MeSH Terms: conditions — Arthritis; Tendinopathy; Gout; Radiculopathy; Spasm; Synovitis; Migraine Disorders; Headache | interventions — Baclofen; Bupivacaine; cyclobenzaprine; Diclofenac; Flurbiprofen; Gabapentin; Ketamine; Lidocaine; Prilocaine; Meloxicam; Sumatriptan; tizanidine; Topiramate; Capsaicin; Menthol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: baclofen 2% — compound topical cream
  Other Names: baclofen
Drug: Bupivacaine hydrochloride 1% — compound topical cream
  Other Names: Bupivacaine hydrochloride
Drug: Cyclobenzaprine hydrochloride 2% — compound topical cream
  Other Names: Cyclobenzaprine hydrochloride
Drug: Diclofenac Sodium 3% — compound topical cream
  Other Names: Diclofenac Sodium
Drug: Flurbiprofen 10% — compound topical cream
  Other Names: Flurbiprofen
Drug: Gabapentin 6% — compound topical cream
  Other Names: Gabapentin
Drug: Ketamine 10% — compound topical cream
  Other Names: Ketamine
Drug: Lidocaine 2% — compound topical cream
  Other Names: Lidocaine
Drug: Prilocaine 2.5% — compound topical cream
  Other Names: Prilocaine
Drug: Meloxicam 0.09% — compound topical cream
  Other Names: Meloxicam
Drug: Sumatriptan 5% — compound topical cream
  Other Names: Sumatriptan
Drug: Tizanidine 0.1% — compound topical cream
  Other Names: Tizanidine
Drug: Topiramate 2.5% — compound topical cream
  Other Names: Topiramate
Drug: Capsaicin, USP 0.0375% — compound topical cream
  Other Names: Capsaicin
Drug: Menthol, NF 5.00 % — compound topical cream
  Other Names: Menthol

SUMMARY:
A 24-week observational prospective study on the efficacy of topical non-steroidal anti-inflammatory drugs for the relief of pain.

DETAILED DESCRIPTION:
Objectives

The primary objective is the change in pain levels as measured by a 10-point visual analog scale (VAS). Secondary objectives are changes in concomitant pain medication use, quality of life, and patient satisfaction with pain management.

Design and Outcomes

The study will be conducted at 1 family practice medical clinic in Houston, TX. Patients will be prescribed a pain cream compound based on their symptoms and medical history. Periodic surveys will be administered and concomitant medications recorded to ascertain current pain levels, quality of life, and satisfaction with current pain levels. Blood tests will be performed to monitor liver and kidney function.

Interventions and Duration

Non-steroidal anti-inflammatory steroid (NSAID) topical cream will be prescribed to patients presenting with pain. For patients with localized pain, they will also be prescribed a transdermal analgesic patch to wear at the site of pain. Subjects will be followed for 24-weeks with surveys administered at baseline, and 1, 2, 4, 8, 12, 16, 20, and 24-weeks after baseline with blood tests performed at 12 and 24-weeks. If patients do not find satisfactory pain relief or experience undesirable side effects from the cream they will be given a prescription for an oral NSAID at anytime during the 24-week observation.

Sample Size and Population

500 patients will be enrolled in the study between March 1, 2015 and March 1, 2017. Subjects will be screened from the patient population at 1960 Family Practice, 837 Cupress Creek Parkway, Suite 105, Houston Texas. Subjects will have presented with a primary complaint of pain. Subjects will be stratified by the following medical indications; Arthritis Muscle Spasms Tendonitis Idiopathic Gout Synovitis Radiculopathy Migraine

ELIGIBILITY:
Inclusion Criteria:

* 4.1.1 Primary complaint or clinical findings of arthritis, tendonitis, gout, synovitis, radiculopathy, muscle spasms, migraines, and/or idiopathic pain.

4.1.2 No new pain medications of any kind in the last 4 weeks. 4.1.3 Between the ages of 18-85yrs.

Exclusion Criteria:

* 4.2.1 Current or history of disease or disorders of the liver, kidneys, gastrointestinal system, or cardiovascular system.

4.2.2 Blood test indicating kidney, liver, or cardiovascular function outside of normal clinically accepted ranges. Blood test must be performed in the last 7 days.

4.2.3 Broken or inflamed skin, burns, open wounds, atopic dermatitis or eczema in the area of pain where the compound cream and transdermal patch would be applied.

4.2.4 Women who are pregnant, nursing, or planning to become pregnant in the next 52-weeks.

4.2.5 Allergy/sensitivity to study drugs or their formulations. 4.2.6 Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

4.2.7 Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 14 days prior to study entry.

4.2.8 Inability or unwillingness of subject to give written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will be taken from the patients normally treated at 1960 Family Practice. Patients not approached for the study will have known medical issues consistent with the exclusion criteria. Patients who can meet the medical requirements of the inclusion criteria for the study will be asked to participate. Patients who do not meet the inclusion criteria, meet any of the exclusion criteria, or decline to be involved in the study will be treated with traditional standard medical practices, and their standard of care will not change in any way.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
subjective pain control as measured by a 10-point visual analog scale (VAS). | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kate McLellan, PhD, Study Director — KM Clinical, Inc.

IPD SHARING:
Plan to Share IPD: No